CLINICAL TRIAL: NCT04285684
Title: The Pharmacokinetics of Ketamine in the Breast Milk of Lactating Women: Quantification of Ketamine and Metabolites
Brief Title: The Pharmacokinetics of Ketamine in the Breast Milk of Lactating Women
Acronym: KRF-LAC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Ketamine Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KetamineResearch
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Results first posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-10

CONDITIONS: Ketamine; Lactation
Keywords: ketamine; lactation; postpartum depression; breastfeeding; infant exposure
MeSH Terms: conditions — Breast Feeding; Depression, Postpartum | interventions — Ketamine; Lactation

STUDY DESIGN:
Intervention Model Description: 4 subjects receiving 0.5mg/kg and 1.0mg/kg of ketamine at least 5 days apart with collection of breast milk by pumping at 3 hour intervals
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine, lactation (Other): Lactating women--4 subjects, 2 dosage format: ketamine 0;5mg/kg and 1.0mg/kg IM at least 5 days apart.
  Interventions: Drug: ketamine in lactation

INTERVENTIONS:
Drug: ketamine in lactation — 2 dose IM by weight and assessing concentrations of ketamine in expressed milk at intervals
  Other Names: Assessing concentration of ketamine in breast milk at intervals

SUMMARY:
Quantification of Ketamine in Breast Milk at 3 hour Intervals up to 30 hours-- obtained from lactating women who receive 2 different Intramuscular injections of ketamine on two separate days at least 5 days apart.

DETAILED DESCRIPTION:
Quantification of Ketamine in Breast Milk at 3 hour Intervals up to 30 hours-- obtained from lactating women who receive 2 different Intramuscular injections of ketamine on two separate days at least 5 days apart: 0.5mg/kg and 1.0mg kg.

Women are required to have been breast feeding for at least 3 months and be healthy and on no medications. Support is provided for the entire time at the site and for any at home pumping. During the period of ketamine's influence, subjects are reclining and with 2 Investigators. The initial subject's data will determine the length of time for pumping--most likely 12 hours as ketamine and the active principle metabolite have half-lives of less than 3 hours. Determination of concentration of ketamine in breast milk is being done at the UCSF Clinical lab with quantification of metabolites that are inactive as well. This research is of benefit by providing lactating women information on potential exposure of infants/children to ketamine. It will serve as a guide as KRF conducts research on postpartum depression and for women at large using ketamine for psychiatric indications.

ELIGIBILITY:
Inclusion Criteria:• Age 21-45

* Postpartum with established lactation for a minimum of 3 months.
* Ability to pump breast milk and to provide a reservoir for infant feeding prior to the study; or acceptance of bottle feeding by the infant.
* In good health-normal BP/P; afebrile-temp ascertained; review of systems by MD; absence of diagnosed illnesses.
* Not pregnant--Pregnancy tested for before each administration by urine assay.

Exclusion Criteria:• Hypertension with a BP greater than 145/90

* Subjects must be off all psychiatric medications specifically; medications and supplements, or evaluated by the PI for non-interference
* No alcohol or other substances such as marijuana for 72 hours or more.
* Weight <50kg or > 90kg.
* Pregnancy

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 4 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Wolfson, MD, Principal Investigator — Ketamine Research Foundation
Locations (1):
- Ketamine Research Foundation, San Anselmo, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication of data in peer reviewed journal including all data; and available from KRF by request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months to 1 year
Access Criteria: Public and researchers Health care professionals
URL: http://www.ketamineresearchfoundation.com

REFERENCES:
- [Background] Chang T, Glazko AJ. Biotransformation and disposition of ketamine. Int Anesthesiol Clin. 1974 Summer;12(2):157-77. doi: 10.1097/00004311-197412020-00018. No abstract available. PMID 4603048
- [Background] Clements JA, Nimmo WS, Grant IS. Bioavailability, pharmacokinetics, and analgesic activity of ketamine in humans. J Pharm Sci. 1982 May;71(5):539-42. doi: 10.1002/jps.2600710516. PMID 7097501
- [Background] Dore J, Turnipseed B, Dwyer S, Turnipseed A, Andries J, Ascani G, Monnette C, Huidekoper A, Strauss N, Wolfson P. Ketamine Assisted Psychotherapy (KAP): Patient Demographics, Clinical Data and Outcomes in Three Large Practices Administering Ketamine with Psychotherapy. J Psychoactive Drugs. 2019 Apr-Jun;51(2):189-198. doi: 10.1080/02791072.2019.1587556. Epub 2019 Mar 27. PMID 30917760
- [Background] Little B, Chang T, Chucot L, Dill WA, Enrile LL, Glazko AJ, Jassani M, Kretchmer H, Sweet AY. Study of ketamine as an obstetric anesthetic agent. Am J Obstet Gynecol. 1972 May 15;113(2):247-60. doi: 10.1016/0002-9378(72)90774-0. No abstract available. PMID 4554554
- [Background] Wan LB, Levitch CF, Perez AM, Brallier JW, Iosifescu DV, Chang LC, Foulkes A, Mathew SJ, Charney DS, Murrough JW. Ketamine safety and tolerability in clinical trials for treatment-resistant depression. J Clin Psychiatry. 2015 Mar;76(3):247-52. doi: 10.4088/JCP.13m08852. PMID 25271445
- [Background] Weber F, Wulf H, Gruber M, Biallas R. S-ketamine and s-norketamine plasma concentrations after nasal and i.v. administration in anesthetized children. Paediatr Anaesth. 2004 Dec;14(12):983-8. doi: 10.1111/j.1460-9592.2004.01358.x. PMID 15601346

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine During Lactation: Participants received 2 ketamine administrations, 0.5mg/kg and 1.0mg/kg IM, at least 5 days apart.
Period: Overall Study
Arm/Group | Ketamine During Lactation
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine During Lactation
Number analyzed (Participants) | 4
Age, Customized [Count of Participants; unit: Participants]
  Between 21 and 45 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 4
Postpartum with Established Lactation for a Minimum of 3 Months [Count of Participants; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: Ketamine Concentration in Breast Milk, up to 12 Hours at 3 Hour Intervals, Following an IM Administration of .5mg/kg Ketamine
Description: Quantitative analysis of the concentration of ketamine and its metabolites in breast milk (collected by pumping breast milk into containers at 3, 6, 9, and 12 hours post ketamine IM administration) was performed at the Clinical Medicine and Toxicology Laboratory at UCSF School of Medicine. Sample aliquots were frozen in our conventional freezer at the clinic where the sessions took place, labelled with a HIPAA compliant code which blinded the lab to all patient data.
  The limits of sensitivity for the quantification of each substance were:
  Ketamine: 0.25 ng Norketamine: 0.25 ng Dehydronorketamine: 0.1 ng Hydroxynorketamine: 0.25 ng
Time Frame: 3, 6, 9, and 12 hour collections
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Ketamine During Lactation: Participants received .5mg/kg and 1mg/kg IM ketamine, at least 5 days apart
Arm/Group | Ketamine During Lactation
Number analyzed (Participants) | 4
ng/mL
  3 Hours | 51.2 (18.8)
  6 Hours | 22.6 (8.4)
  9 Hours | 10.6 (5.4)
  12 Hours | 4.5 (4.4)

2. Primary Outcome: Ketamine Concentration in Breast Milk, up to 12 Hours at 3 Hour Intervals, Following an IM Administration of 1mg/kg Ketamine
Description: as for outcome 1
Time Frame: 3, 6, 9, and 12 hour collections
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketamine During Lactation
Number analyzed (Participants) | 4
ng/mL
  3 Hours | 125.0 (44.1)
  6 Hours | 48.2 (17.3)
  9 Hours | 21.6 (13.9)
  12 Hours | 18.5 (6.7)

3. Primary Outcome: Norketamine Concentration in Breast Milk, up to 12 Hours at 3 Hour Intervals, Following an IM Administration of .5mg/kg Ketamine
Description: as for outcome 1
Time Frame: 3, 6, 9, and 12 hour collections
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketamine During Lactation
Number analyzed (Participants) | 4
ng/mL
  3 Hours | 42.6 (10.5)
  6 Hours | 28.6 (5.2)
  9 Hours | 18.8 (5.1)
  12 Hours | 8.7 (6.4)

4. Primary Outcome: Norketamine Concentration in Breast Milk, up to 12 Hours at 3 Hour Intervals, Following an IM Administration of 1mg/kg Ketamine
Description: as for outcome 1
Time Frame: 3, 6, 9, and 12 hour collections
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketamine During Lactation
Number analyzed (Participants) | 4
ng/mL
  3 Hours | 92.7 (14.8)
  6 Hours | 62.4 (12.9)
  9 Hours | 37.3 (10.5)
  12 Hours | 32.3 (10.3)

5. Primary Outcome: Dehydronorketamine Concentration in Breast Milk, up to 12 Hours at 3 Hour Intervals, Following an IM Administration of .5mg/kg Ketamine
Description: as for outcome 1
Time Frame: 3, 6, 9, and 12 hour collections
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketamine During Lactation
Number analyzed (Participants) | 4
ng/mL
  3 Hours | .56 (.3)
  6 Hours | .55 (.2)
  9 Hours | .45 (.3)
  12 Hours | .21 (.1)

6. Primary Outcome: Dehydronorketamine Concentration in Breast Milk, up to 12 Hours at 3 Hour Intervals, Following an IM Administration of 1mg/kg Ketamine
Description: as for outcome 1
Time Frame: 3, 6, 9, and 12 hour collections
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketamine During Lactation
Number analyzed (Participants) | 4
ng/mL
  3 Hours | 2.0 (1.1)
  6 Hours | 1.9 (1.1)
  9 Hours | 1.4 (.7)
  12 Hours | 1.1 (.7)

7. Primary Outcome: Hydroxynorketamine Concentration in Breast Milk, up to 12 Hours at 3 Hour Intervals, Following an IM Administration of .5mg/kg Ketamine
Description: as for outcome 1
Time Frame: 3, 6, 9, and 12 hour collections
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketamine During Lactation
Number analyzed (Participants) | 4
ng/mL
  3 Hours | 29.9 (9.0)
  6 Hours | 28.3 (10.2)
  9 Hours | 25.6 (8.0)
  12 Hours | 17.5 (9.9)

8. Primary Outcome: Hydroxynorketamine Concentration in Breast Milk, up to 12 Hours at 3 Hour Intervals, Following an IM Administration of 1mg/kg Ketamine
Description: as for outcome 1
Time Frame: 3, 6, 9, and 12 hour collections
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketamine During Lactation
Number analyzed (Participants) | 4
ng/mL
  3 Hours | 64.1 (21.1)
  6 Hours | 66.9 (13.1)
  9 Hours | 54.6 (11.2)
  12 Hours | 41.6 (9.8)

9. Primary Outcome: Ketamine Concentration in Breast Milk at 24 and 30 Hours After an IM Administration of 1mg/kg Ketamine
Description: Quantitative analysis of the concentration of ketamine and its metabolites in breast milk (collected by pumping breast milk into containers at 24 and 30 hours post ketamine IM administration) was performed at the Clinical Medicine and Toxicology Laboratory at UCSF School of Medicine. Sample aliquots were frozen in our conventional freezer at the clinic where the sessions took place, labelled with a HIPAA compliant code which blinded the lab to all patient data.
  The limits of sensitivity for the quantification of each substance were:
  Ketamine: 0.25 ng Norketamine: 0.25 ng Dehydronorketamine: 0.1 ng Hydroxynorketamine: 0.25 ng
Time Frame: 24 and 30 hour collections
Population: Based on the concentration of ketamine and its metabolites at 24 and 30 hours post ketamine administration in the first participant tested, breast milk was not collected for subsequent participants at these time frames.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketamine During Lactation
Number analyzed (Participants) | 1
ng/mL
  24 Hours | 4.9 (NA) — Standard Deviation is not calculable for one participant.
  30 Hours | 6.4 (NA) — Standard Deviation is not calculable for one participant.

10. Primary Outcome: Norketamine Concentration in Breast Milk at 24 and 30 Hours After an IM Administration of 1mg/kg Ketamine
Description: as for outcome 9
Time Frame: 24 and 30 hour collections
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketamine During Lactation
Number analyzed (Participants) | 1
ng/mL
  24 Hours | 10.3 (NA) — Standard Deviation is not calculable for one participant.
  30 Hours | 9.9 (NA) — Standard Deviation is not calculable for one participant.

11. Primary Outcome: Dehydronorketamine Concentration in Breast Milk at 24 and 30 Hours After an IM Administration of 1mg/kg Ketamine
Description: as for outcome 9
Time Frame: 24 and 30 hour collections
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketamine During Lactation
Number analyzed (Participants) | 1
ng/mL
  24 Hours | .3 (NA) — Standard Deviation is not calculable for one participant.
  30 Hours | .3 (NA) — Standard Deviation is not calculable for one participant.

12. Primary Outcome: Hydroxynorketamine Concentration in Breast Milk at 24 and 30 Hours After an IM Administration of 1mg/kg Ketamine
Description: as for outcome 9
Time Frame: 24 and 30 hour collections
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketamine During Lactation
Number analyzed (Participants) | 1
ng/mL
  24 Hours | 30.5 (NA) — Standard Deviation is not calculable for one participant.
  30 Hours | 13.9 (NA) — Standard Deviation is not calculable for one participant.

ADVERSE EVENTS:
Time Frame: Adverse event data was collected continuously starting with the first ketamine administration, through the second ketamine administration (5-14 days following the first administration), and during a formal four week follow-up thereafter.
Arm/Group | Ketamine During Lactation
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
After the collection of breast milk from the first subject, it was determined that 3 hour intervals up to 12 hours was a sufficient collection period for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT04285684/Prot_SAP_000.pdf